## **Clinical Research Abstract**

| Brief Title Study on the Correlation Between Treg Immune Cells on the Muscle Content and Cognitive Functions of the Elderly ID ZDWY.LNBK.007 Sponsor Fifth Affiliated Hospital, Sun Yat-Sen University Research unit Main researcher Statistical unit and person in charge of statistics In order to explore the impact of the level of the elderly TREG immune cells and the effects of different fat distribution and muscle content, the impact of the level of TREG immune cells and cognitive function. Sample size Selected standards For subjects Research step Accelerated Standards For subjects Research step Accelerated Standards Bresearch step 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The impact of the level of TREG immune cells on cognitive function; 4. | | |
|---|---|---|
| Content and Cognitive Functions of the Elderly | Brief Title | Study on the Correlation Between Treg Immune Cells on the Muscle |
| Research unit Fifth Affiliated Hospital, Sun Yat-Sen University | | Content and Cognitive Functions of the Elderly |
| Research unit Main researcher Wenya Han Fifth Affiliated Hospital, Sun Yat-Sen University Wenya Han Fifth Affiliated Hospital, Sun Yat-Sen University Wenya Han Fith Affiliated Hospital Fusion Fusion Table Place Indicates Fusion Table Place Indicate | ID | ZDWY.LNBK.007 |
| Statistical unit and person in charge of statistics | Sponsor | Fifth Affiliated Hospital, Sun Yat-Sen University |
| Statistical unit and person in charge of statistics In order to explore the impact of the level of the elderly TREG immune cells and the effects of different fat distribution and muscle content, the impact of the level of TREG immune cells on cognitive functions is explored. The correlation between visceral fat content, subcutaneous fat content and cognitive function. Sample size 100 Study Type Observational Inclusion criteria: 1. 40-90 years old Exclusion criteria: previous diagnosis of dementia (including Alzheimer's disease, Lewy body dementia, Parkinson's disease, or other dementias) were excluded. 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | Research unit | Fifth Affiliated Hospital, Sun Yat-Sen University |
| Research purposes In order to explore the impact of the level of the elderly TREG immune cells and the effects of different fat distribution and muscle content, the impact of the level of TREG immune cells on cognitive functions is explored. The correlation between visceral fat content, subcutaneous fat content and cognitive function. Sample size 100 Study Type Observational Inclusion criteria: 1. 40-90 years old Exclusion criteria: previous diagnosis of dementia (including Alzheimer's disease, Lewy body dementia, Parkinson's disease, or other dementias) were excluded. 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | Main researcher | Wenya Han |
| In order to explore the impact of the level of the elderly TREG immune cells and the effects of different fat distribution and muscle content, the impact of the level of TREG immune cells on cognitive functions is explored. The correlation between visceral fat content, subcutaneous fat content and cognitive function. Sample size 100 Study Type Observational Inclusion criteria: 1. 40-90 years old Exclusion criteria: previous diagnosis of dementia (including Alzheimer's disease, Lewy body dementia, Parkinson's disease, or other dementias) were excluded. 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | Statistical unit and | Fifth Affiliated Hospital, Sun Yat-Sen University Wenya Han |
| In order to explore the impact of the level of the elderly TREG immune cells and the effects of different fat distribution and muscle content, the impact of the level of TREG immune cells on cognitive functions is explored. The correlation between visceral fat content, subcutaneous fat content and cognitive function. Sample size | person in charge of | |
| cells and the effects of different fat distribution and muscle content, the impact of the level of TREG immune cells on cognitive functions is explored. The correlation between visceral fat content, subcutaneous fat content and cognitive function. Sample size 100 Study Type Observational Inclusion criteria: 1. 40-90 years old Exclusion criteria: previous diagnosis of dementia (including Alzheimer's disease, Lewy body dementia, Parkinson's disease, or other dementias) were excluded. 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | statistics | |
| Research purposes impact of the level of TREG immune cells on cognitive functions is explored. The correlation between visceral fat content, subcutaneous fat content and cognitive function. Sample size 100 Study Type Observational Inclusion criteria: 1. 40-90 years old Exclusion criteria: previous diagnosis of dementia (including Alzheimer's disease, Lewy body dementia, Parkinson's disease, or other dementias) were excluded. 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | | In order to explore the impact of the level of the elderly TREG immune |
| explored. The correlation between visceral fat content, subcutaneous fat content and cognitive function. Sample size 100 Study Type Observational Inclusion criteria: 1. 40-90 years old Exclusion criteria: previous diagnosis of dementia (including Alzheimer's disease, Lewy body dementia, Parkinson's disease, or other dementias) were excluded. 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | | cells and the effects of different fat distribution and muscle content, the |
| content and cognitive function. Sample size 100 Study Type Observational Inclusion criteria: 1. 40-90 years old Exclusion criteria: previous diagnosis of dementia (including Alzheimer's disease, Lewy body dementia, Parkinson's disease, or other dementias) were excluded. 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | Research purposes | impact of the level of TREG immune cells on cognitive functions is |
| Study Type Observational Inclusion criteria: 1. 40-90 years old Exclusion criteria: previous diagnosis of dementia (including Alzheimer's disease, Lewy body dementia, Parkinson's disease, or other dementias) were excluded. 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | | explored. The correlation between visceral fat content, subcutaneous fat |
| Selected standards for subjects Selected standards 1. 40-90 years old | | content and cognitive function. |
| Inclusion criteria: 1. 40-90 years old | Sample size | 100 |
| 1. 40-90 years old Exclusion criteria: previous diagnosis of dementia (including Alzheimer's disease, Lewy body dementia, Parkinson's disease, or other dementias) were excluded. 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | Study Type | Observational |
| For subjects previous diagnosis of dementia (including Alzheimer's disease, Lewy body dementia, Parkinson's disease, or other dementias) were excluded. 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | | Inclusion criteria: |
| previous diagnosis of dementia (including Alzheimer's disease, Lewy body dementia, Parkinson's disease, or other dementias) were excluded. 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | | 1. 40-90 years old |
| body dementia, Parkinson's disease, or other dementias) were excluded. 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | Selected standards | Exclusion criteria: |
| excluded. 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | for subjects | previous diagnosis of dementia (including Alzheimer's disease, Lewy |
| 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting in our hospital at the same time improve the data measurement and TREG cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | | body dementia, Parkinson's disease, or other dementias) were |
| in our hospital at the same time improve the data measurement and TREG Research step cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | | excluded. |
| Research step cell measurement data at the same time; 2. The level of TREG immune cells and different fat distribution and muscle content Impact; 3. The | | 1. Collect 2023-05-01 to 2024-12-31 Elderly patients who are consulting |
| cells and different fat distribution and muscle content Impact; 3. The | | in our hospital at the same time improve the data measurement and TREG |
| | Research step | cell measurement data at the same time; 2. The level of TREG immune |
| impact of the level of TREG immune cells on cognitive function; 4. | | cells and different fat distribution and muscle content Impact; 3. The |
| | | impact of the level of TREG immune cells on cognitive function; 4. |

| | Evaluate the effects of different fat distribution and muscle content on |
|---|---|
| | cognitive functions, evaluate the correlation between internal organs, |
| | subcutaneous fat content and cognitive functions; 5. Write the paper. |
| Terminal indicator | Cognitive function decline |
| | Use a linear regression model to analyze the level of the level of TREG |
| | immune cells, the effects of different fat distribution and muscle content; |
| | the impact of the level of TREG immune cells on the level of TREG |
| | immune cells is analyzed by the Mann-Whitney U test; the evaluation of |
| Statistical Analysis | different fat distribution and muscle content The impact on cognitive |
| | functions, evaluate the correlation between the content of visceral fat, |
| | subcutaneous fat content and cognitive functions. |
| | Statistical software includes SPSS27 and Graphpad Prism 8. Inspection |
| | level $\alpha = 0.05$ . |